CLINICAL TRIAL: NCT00278785
Title: Brief Intervention for Alcohol Use Among Injured Patients: A Prospective, Randomized Trial
Brief Title: Brief Intervention for Alcohol Use Among Injured Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Office of Traffic Safety (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 237217; Office of Traffic Safety (Other: UC Davis); Grant Number AL0584 (Other Grant/Funding Number: UC Davis)
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Drinking; Wounds and Injuries
Keywords: interviews; brief intervention; drinking; alcohol; injuries; wounds; intervention studies
MeSH Terms: conditions — Alcohol Drinking; Wounds and Injuries | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control group to receive informational pamphlet on alcohol use and list of self referral agencies
- 2 (Experimental): Intervention group receives pamphlet on alcohol and self referral information in addition to brief motivational interview
  Interventions: Behavioral: Brief Motivational Interview

INTERVENTIONS:
Behavioral: Brief Motivational Interview — 10-20 minute brief motivational interview
  Other Names: Brief intervention; Motivational interview
  Arms: 2

SUMMARY:
The underlying hypothesis that providing brief interventions to individuals who engage in potentially harmful patterns of alcohol use will alter their drinking behavior and therefore avoid negative consequences. Specifically, this study aims to determine if brief interventions will:

1. Reduce the number of re-admissions and deaths due to injuries associated with alcohol consumption
2. Reduce the number of driving under the influence (DUI) arrests
3. Reduce harmful drinking behavior

DETAILED DESCRIPTION:
Alcohol use is the most common underlying cause of injuries in the United States. There is a growing body of literature suggesting that brief interventions (BI), in the form of a short (10-60 minute) counseling session, may decrease alcohol consumption and its harmful consequences. In contrast to the abundant literature on the effectiveness of BI in the outpatient setting, only 3 randomized controlled trials have been performed an adults specifically in the setting of acute trauma, and have had inconclusive results. All three studies used highly trained persons to perform the BI, and all were greater than 30 minutes in duration, a situation that may not necessarily reflect the practicalities of routine medical care. This raises the question of whether the benefits seen in these studies reflect the expertise of a small number of individuals or whether the effects correlate with the amount of time spent with the patient. Highly trained personnel and time are valuable commodities in a busy trauma center and may not be feasible given the competing clinical demands. We propose to investigate whether BI are effective in a setting that is more likely to reflect "real world" of clinical medicine rather than an idealized setting, utilizing trauma nurse practitioners to perform brief (5-10 minute) interviews.

We will identify all patients admitted with trauma who test positive on a blood alcohol test. These patients will be consented and randomized to either a brief intervention group, or a standard medical care group. All patients will receive an AUDIT questionnaire to identify patterns of drinking behavior and an alcohol information pamphlet. After discharge, patients will be telephoned at 1,6, and 12 months. The first 2 contacts will be to see how the patient is doing and to verify the contact information. The AUDIT questionnaire will be re-administered during the 12 month interview.

ELIGIBILITY:
Inclusion Criteria:

* >=18 yrs old
* English or Spanish Speaking
* Mentally and physically able to provide consent and participate in the intervention
* Admission to the trauma ward or ICU

Exclusion Criteria:

* <18 yrs old
* Non-English or Non-Spanish Speaking
* Severe Psychiatric illness
* incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2006-03; Primary Completion 2027-01-24 (Estimated); Study Completion 2027-01-24 (Estimated)

PRIMARY OUTCOMES:
Hospital re-admissions | 2 years
  number of hospital re-admissions

SECONDARY OUTCOMES:
12 month AUDIT Results | 12 months
  Score on self administered questionnaire
Moving violations/DUI | 2 years
  number of moving violations/DUI
Self referral for counselling/treatment | 12 months
  number of self referrals for counseling/treatment

CONTACTS AND LOCATIONS:
Overall Officials: Garth H. Utter, MD, MSc, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Gentilello LM, Donovan DM, Dunn CW, Rivara FP. Alcohol interventions in trauma centers. Current practice and future directions. JAMA. 1995 Oct 4;274(13):1043-8. PMID 7563455
- [Background] Soderstrom CA, Smith GS, Dischinger PC, McDuff DR, Hebel JR, Gorelick DA, Kerns TJ, Ho SM, Read KM. Psychoactive substance use disorders among seriously injured trauma center patients. JAMA. 1997 Jun 11;277(22):1769-74. PMID 9178789
- [Background] Rivara FP, Koepsell TD, Jurkovich GJ, Gurney JG, Soderberg R. The effects of alcohol abuse on readmission for trauma. JAMA. 1993 Oct 27;270(16):1962-4. PMID 8105114
- [Background] Gentilello LM, Rivara FP, Donovan DM, Jurkovich GJ, Daranciang E, Dunn CW, Villaveces A, Copass M, Ries RR. Alcohol interventions in a trauma center as a means of reducing the risk of injury recurrence. Ann Surg. 1999 Oct;230(4):473-80; discussion 480-3. doi: 10.1097/00000658-199910000-00003. PMID 10522717
- [Background] Ockene JK, Adams A, Hurley TG, Wheeler EV, Hebert JR. Brief physician- and nurse practitioner-delivered counseling for high-risk drinkers: does it work? Arch Intern Med. 1999 Oct 11;159(18):2198-205. doi: 10.1001/archinte.159.18.2198. PMID 10527297
- [Background] Smith AJ, Hodgson RJ, Bridgeman K, Shepherd JP. A randomized controlled trial of a brief intervention after alcohol-related facial injury. Addiction. 2003 Jan;98(1):43-52. doi: 10.1046/j.1360-0443.2003.00251.x. PMID 12492754
- [Background] Spirito A, Monti PM, Barnett NP, Colby SM, Sindelar H, Rohsenow DJ, Lewander W, Myers M. A randomized clinical trial of a brief motivational intervention for alcohol-positive adolescents treated in an emergency department. J Pediatr. 2004 Sep;145(3):396-402. doi: 10.1016/j.jpeds.2004.04.057. PMID 15343198
- [Background] Monti PM, Colby SM, Barnett NP, Spirito A, Rohsenow DJ, Myers M, Woolard R, Lewander W. Brief intervention for harm reduction with alcohol-positive older adolescents in a hospital emergency department. J Consult Clin Psychol. 1999 Dec;67(6):989-94. doi: 10.1037//0022-006x.67.6.989. PMID 10596521
- [Background] Longabaugh R, Woolard RE, Nirenberg TD, Minugh AP, Becker B, Clifford PR, Carty K, Licsw, Sparadeo F, Gogineni A. Evaluating the effects of a brief motivational intervention for injured drinkers in the emergency department. J Stud Alcohol. 2001 Nov;62(6):806-16. doi: 10.15288/jsa.2001.62.806. PMID 11838918